CLINICAL TRIAL: NCT00329251
Title: Study of the Influence of Immunological Repeated Stimuli With Commercial Vaccines Over the Viral Load (VL), Resistance Development and Specific Immunological Response Against HIV in Early Stage HIV Patients With Undetectable VL After HAART
Brief Title: Study of the Influence of Vaccination in HIV Viral Load and Immunologic Responses Against HIV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02-0490; EARTH-06; VAC-01
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2006-05-24 (Estimated); Status verified 2006-05

CONDITIONS: HIV
Keywords: HIV; Viral load; Vaccines; Immunotherapy
MeSH Terms: interventions — Hepatitis A Vaccines; Hepatitis B Vaccines; Influenza Vaccines

INTERVENTIONS:
Biological: Hepatitis A
Biological: Hepatitis B
Biological: Influenza
Biological: Pneumococcal
Biological: Tetanus-diphteria
Biological: Varicella
Biological: Measles-Mumps-Rubella

SUMMARY:
The purpose of this study is to determine whether an immunization schedule is beneficial to HIV-infected patients with CD4 recount over 500 cells/mm3 and undetectable viral load.

DETAILED DESCRIPTION:
As HIV-infected patients are considered immunocompromised, it is generally recommended that they have to receipt appropriate vaccines. However data are conflicting concerning potential harmful effects following the administration of commercial vaccines in HIV-infected patients. Transient increases ("blips") in the viral load have been described associated with a single dose of vaccine, with the potential risk of developing resistance to HAART. On the other hand, there has been described that patients with blips can have an increase in HIV-specific immune responses, which may help to improve the viral control.

Comparison: We have performed a clinical trial to evaluate the effect of a vaccination program in successfully treated HIV-infected adults on HAART compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Asymptomatic HIV infection
* CD4>500/mm3 >6 months prior to inclusion
* CD4 nadir >300/mm3
* Being under HAART > 1 year prior to inclusion
* Viral load<200 copies/mL > 6 months prior to inclusion
* Viral load previous to treatment >5000 copies/mL
* Informed consent

Exclusion Criteria:

* Pregnant women
* Basal creatinine >2.5 mg/dL
* Allergy to either a vaccine or a ingredient of it
* Chronic hepatitis B
* GOT/GPT > 250 IU/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26
Dates: Start 2003-04; Study Completion 2006-03

PRIMARY OUTCOMES:
Times viral load increases over 20.000 copies/mL.

SECONDARY OUTCOMES:
Development of resistance to antiretroviral therapy during the 18 months of the study
Appearance of specific CD4 proliferative responses against HIV during the 18 months of the study
Appearance of specific cytotoxic responses against HIV during the 18 months of the study
Number of patients under 5000 copies/mL after 6 months of stopping HAART
Development of symptoms C during the 18 months of the study
Deaths during the 18 months of the study
Toxicity during the 18 months of the study

CONTACTS AND LOCATIONS:
Overall Officials: José Mª Gatell, MD, Study Chair — Hospital Clínic of Barcelona; José Mª Miró, MD, Study Chair — Hospital Clínic of Barcelona; José Mª Bayas, MD, Study Chair — Hospital Clínic of Barcelona
Locations (1):
- Department of Infectious Diseases, Hospital Clínic, C/Villarroel 170, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Yek C, Gianella S, Plana M, Castro P, Scheffler K, Garcia F, Massanella M, Smith DM. Standard vaccines increase HIV-1 transcription during antiretroviral therapy. AIDS. 2016 Sep 24;30(15):2289-98. doi: 10.1097/QAD.0000000000001201. PMID 27427877
- [Derived] Castro P, Torres B, Lopez A, Gonzalez R, Vilella A, Nicolas JM, Gallart T, Pumarola T, Sanchez M, Leal M, Vallejo A, Bayas JM, Gatell JM, Plana M, Garcia F. Effects of different antigenic stimuli on thymic function and interleukin-7/CD127 system in patients with chronic HIV infection. J Acquir Immune Defic Syndr. 2014 Aug 15;66(5):466-72. doi: 10.1097/QAI.0000000000000207. PMID 24820104
- [Derived] Castro P, Plana M, Gonzalez R, Lopez A, Vilella A, Nicolas JM, Gallart T, Pumarola T, Bayas JM, Gatell JM, Garcia F. Influence of episodes of intermittent viremia ("blips") on immune responses and viral load rebound in successfully treated HIV-infected patients. AIDS Res Hum Retroviruses. 2013 Jan;29(1):68-76. doi: 10.1089/AID.2012.0145. Epub 2012 Dec 16. PMID 23121249